CLINICAL TRIAL: NCT02981862
Title: Monocentric Study of Validation of the Method "CaptHPV" for the Diagnosis of Human Papillomavirus Associated Infiltrating Carcinomas From a Biological Specimen.
Brief Title: CaptHPV : Validation of the Method "CaptHPV" for the Diagnosis of Human Papillomavirus Associated Infiltrating Carcinomas
Acronym: CaptHPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A01085-46
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Cervical Cancer; Vulvar Cancer; Anal Cancer; Oropharynx Cancer; Oral Cavity Cancer; Penis Cancer
Keywords: HPV infection; Blood sample; Biopsy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Anus Neoplasms; Oropharyngeal Neoplasms; Mouth Neoplasms; Penile Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CaptHPV method (Experimental)
  Interventions: Other: CaptHPV method

INTERVENTIONS:
Other: CaptHPV method — 20 ml of blood sample will be made before the beginning of all treatment. This blood sample will be sent to the CERBA Laboratory for analysis.
  In parallel, a standard anatomopathological and virological analysis will be carried out from a biopsy or from a tumor sample by the Tumor Biology Unit at Lorraine Institute of Oncology
  The results of both analyzes will be compared blindly.

SUMMARY:
The current project is based on the assumption that a diagnosis of human papillomavirus associated Infiltrating Carcinomas can be made from a blood sample for patient with Cervical Cancer, Vulvar Cancer, Anal Cancer, Oropharynx Cancer, Oral Cavity Cancer or Penis Cancer at any stage of the disease and including surgical treatment for the small tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patient with cervical cancer, vulvar cancer, anal cancer, oropharynx cancer, oral cavity cancer or penis cancer
* Patient naive of any treatment for this pathology
* Patient capable and willing to follow all procedures of the study in accordance with the study
* Ability to provide an informed written consent form
* Affiliation to a social security system

Exclusion Criteria:

* Patients who have already undergone surgical treatment leading to complete removal of the lesions or who have started treatment with radiotherapy and / or chemotherapy
* Patient whose health status contraindicates a blood sample of 20 ml,
* Absence of informed written consent form
* Pregnant or breast feeding females
* Patients deprived of liberty or under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Assessement of CaptHPV method | 1 day
  The diagnostic value of the serum marker provided by the method CaptHPV will be assessed in sensitivity and specificity to results of histological and virological analyzes of a sample tumor.

CONTACTS AND LOCATIONS:
Overall Officials: SASTRE-GARAU Xavier, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sastre-Garau X, Diop M, Martin F, Dolivet G, Marchal F, Charra-Brunaud C, Peiffert D, Leufflen L, Dembele B, Demange J, Tosti P, Thomas J, Leroux A, Merlin JL, Diop-Ndiaye H, Costa JM, Salleron J, Harle A. A NGS-based Blood Test For the Diagnosis of Invasive HPV-associated Carcinomas with Extensive Viral Genomic Characterization. Clin Cancer Res. 2021 Oct 1;27(19):5307-5316. doi: 10.1158/1078-0432.CCR-21-0293. PMID 34108183